CLINICAL TRIAL: NCT05933616
Title: Analysis of Volatile Organic Compounds in Patients With Type 1 Diabetes in Induced Hypoglycaemia With a Breath Analyser
Acronym: VAARABreath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: DCB Research AG (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VAARABreath
Record Dates: First submitted 2023-06-26; First posted 2023-07-06 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus; Metabolic Disease; Glucose Metabolism Disorders; Endocrine System Diseases
Keywords: Volatile Organic Compounds; Hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Diseases; Glucose Metabolism Disorders; Endocrine System Diseases; Hypoglycemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Participants in the study arm will undergo the study procedure which are different induced glycaemic states.
  Interventions: Device: Device: Sokru device

INTERVENTIONS:
Device: Device: Sokru device — Different induced glycaemic states in people living with diabetes (PwD).

SUMMARY:
The breath analysis (BreathSpec® device) data of all participants that were included into the VAARA study (NCT05771090) will be analysed, this includes data from up to 40 breath samples from each of the 10 participants who underwent 2 insulin-induced hypoglycaemic episodes during two visits. The primary objective is to find a possible association between volatile organic compounds (VOCs) measured by the BreathSpec® device and blood glucose. For this we will use descriptive statistics, correlation coefficients, as well as a Principal Component Analysis and a partial least squares discriminant analysis. Furthermore, the time lag between hypoglycaemia onset and change in VOCs will be quantified.

ELIGIBILITY:
(as in VAARA study, NCT05771090)

Inclusion Criteria:

* Written informed consent.
* Type 1 Diabetes with Multiple daily insulin injection (MDI) or Continuous subcutaneous insulin infusion therapy (CSII) >1 year
* Age 18 - 50 (inclusive)
* Caucasian ethnicity
* BMI between 18.5 and 24.9 kg/m2 (inclusive)
* Usage of a continuous glucose monitoring (CGM)

Exclusion Criteria:

* Pregnancy or lactation period
* History of cardiovascular diseases
* Diabetes-related comorbidities
* HbA1c >9 %
* Epilepsy
* Smoking (last cigarette within past 6 months)
* Known sensitivity to medical grade adhesives or other skin-related complications, which might influence the outcome.
* Known sensitivity to Latex.
* Participation in another investigation with an investigational drug within the 30 days preceding and during the present investigation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Changes VOC Patterns over time as gallery plots | During the study procedure (approximately 5 hours)
  Difference in gallery plots (3D visualization of retention index, drift time, ion current) from selected VOC peaks over time.
Changes VOC Patterns over time as boxplots | During the study procedure (approximately 5 hours)
  Difference in box plots from selected VOC peaks over time.
Correlation between blood glucose and patterns | During the study procedure (approximately 5 hours)
  Signals will be classified into euglycemic (between 4 and 10 mmol/l), hypoglycaemic (smaller than 4 mmol/l) and hyperglycaemic (above 10 mmol/l) phases or stable and changing phases. A principal component analysis (PCA) of the data will be performed to identify which VOCs are characteristic for certain glucose levels. A partial least squares discriminant analysis (PLS-DA) will be used to further identify important features of the VOC fingerprints.

SECONDARY OUTCOMES:
Time lag | During the study procedure (approximately 5 hours)
  The time lag between hypoglycaemia onset and change in VOCs will be calculated-
Association between the onset of change in glucose, vital signs and VOC spectra | During the study procedure (approximately 5 hours)
  Associations between changes in VOCs and perceived hypoglycaemic symptoms, heart rate, ECG, and oxygen saturation will be evaluated using correlation coefficients and mixed effects models.

CONTACTS AND LOCATIONS:
Overall Officials: Witthauer Lilian, Prof.Dr., Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No